CLINICAL TRIAL: NCT05129033
Title: A Prospective, Two-center, Clinical Study to Optimize the Treatment for Allergic Bronchopulmonary Aspergillosis (ABPA)
Brief Title: A Prospective Study on Optimizing Treatment for ABPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020ZSLC26
Record Dates: First submitted 2021-07-03; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Allergic Bronchopulmonary Aspergillosis
Keywords: Allergic Bronchopulmonary Aspergillosis; anti-fungal agent; Omalizumab; oral corticosteroids
MeSH Terms: conditions — Aspergillosis, Allergic Bronchopulmonary | interventions — Prednisone; Itraconazole; Omalizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-fungal agent plus OCS (Active Comparator): Prednisone tablets is given orally 0.5mg/kg/d for 4 weeks and gradually reduced to stop for a total usage of 6 months Itraconazole is given orally 200mg bid for 8 months and 100mg bid for another 8 months
  Interventions: Drug: Prednisone tablet; Drug: itraconazole
- anti-IgE mAb plus OCS (Active Comparator): Prednisone tablets is given orally 0.5mg/kg/d for 4 weeks and gradually reduced to stop for a total usage of 6 months Omalizumab is given by subcutaneous injection of 600mg q4w for at least 6 months
  Interventions: Drug: Prednisone tablet; Biological: Omalizumab

INTERVENTIONS:
Drug: Prednisone tablet — Basic medication for allergic airway inflammation such as asthma and ABPA, to relieve inflammation. Reduction may failed if disease exacerbate.
Drug: itraconazole — Anti-fungal medication to reduce fugal load.
  Arms: anti-fungal agent plus OCS
Biological: Omalizumab — Anti-IgE monoclonal antibody, used for high IgE allergic disease.
  Arms: anti-IgE mAb plus OCS

SUMMARY:
This study is being done to evaluate the efficacy of treatment using oral glucocorticoid, anti-fungal agent, anti-IgE mAb for patient with ABPA.

DETAILED DESCRIPTION:
This is a study randomly treating ABPA patients with either anti-fungal agent plus OCS or anti-IgE mAb (omalizumab) plus OCS.

OCS is the basic treatment for ABPA by suppressing allergy and inflammation. Prednisone tablets is given orally 0.5mg/kg/d for 4 weeks and gradually reduced to for a total usage of 6 months. Reduction may failed if disease exacerbate.

Anti-fungal agent (mainly itraconazole) could reduce the load of fungus but its application is still controversial. The investigators use itraconazole 200mg bid for 8 months and 100mg bid for another 8 months.

Omalizumab was given 600mg q4w for at least 6 months. The investigators use Anti-fungal agent and Omalizumab as a supplement to OCS to evaluate the better treatment plan for ABPA patients.

ELIGIBILITY:
Inclusion Criteria:

* 18~75 years old, male or female
* associated past medical history, including asthma, bronchiectasis, COPD ect.
* elevated serum total IgE (>100IU/mL)
* elevated aspergillus specific IgE

Exclusion Criteria:

* According to the investigator, the patient has other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, other serious diseases (including mental illness).
* Pregnancy or breastfeeding
* Abnormality of liver or kidney function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-15 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
incidence of exacerbation: the exacerbation times indicated by symptoms and clinical index | Up to 6 months after last treatment dose
  the exacerbation times indicated by symptoms and clinical index, including commom respiratory symptoms such as wheezing, cough, expectation, dyspnea and so on. As well as new shadows in chest CT. Those situation may cause the extreme clinic visit and hospitalization, which could be measured by times or days.

SECONDARY OUTCOMES:
ST.George's respiratory questionnaire | Up to 6 months after last treatment dose
  The SGRQ is a classic respiratory questionnaire including the symptoms, activity, and impact to life. The higher score means better disease control.
asthma control test questionnaire | Up to 6 months after last treatment dose
  The ACT is a classic asthma questionnaire recommended by GINA (Global Initiative for Asthma). ACT mainly measures the symptoms. The higher score means better disease control.

CONTACTS AND LOCATIONS:
Overall Officials: Meiling Jin, MD, Study Chair — Department of Respiratory, Zhongshan Hospital, Fudan University Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agarwal R. Allergic bronchopulmonary aspergillosis. Chest. 2009 Mar;135(3):805-826. doi: 10.1378/chest.08-2586. PMID 19265090
- [Background] Agarwal R, Aggarwal AN, Gupta D, Jindal SK. Aspergillus hypersensitivity and allergic bronchopulmonary aspergillosis in patients with bronchial asthma: systematic review and meta-analysis. Int J Tuberc Lung Dis. 2009 Aug;13(8):936-44. PMID 19723372
- [Background] Agarwal R, Nath A, Aggarwal AN, Gupta D, Chakrabarti A. Aspergillus hypersensitivity and allergic bronchopulmonary aspergillosis in patients with acute severe asthma in a respiratory intensive care unit in North India. Mycoses. 2010 Mar 1;53(2):138-43. doi: 10.1111/j.1439-0507.2008.01680.x. Epub 2009 Jan 24. PMID 19207831
- [Background] Agarwal R, Chakrabarti A, Shah A, Gupta D, Meis JF, Guleria R, Moss R, Denning DW; ABPA complicating asthma ISHAM working group. Allergic bronchopulmonary aspergillosis: review of literature and proposal of new diagnostic and classification criteria. Clin Exp Allergy. 2013 Aug;43(8):850-73. doi: 10.1111/cea.12141. PMID 23889240
- [Background] Mou Y, Ye L, Ye M, Yang D, Jin M. A retrospective study of patients with a delayed diagnosis of allergic bronchopulmonary aspergillosis/allergic bronchopulmonary mycosis. Allergy Asthma Proc. 2014 Mar-Apr;35(2):e21-6. doi: 10.2500/aap.2014.35.3731. PMID 24717781
- [Background] Agarwal R, Gupta D, Aggarwal AN, Saxena AK, Chakrabarti A, Jindal SK. Clinical significance of hyperattenuating mucoid impaction in allergic bronchopulmonary aspergillosis: an analysis of 155 patients. Chest. 2007 Oct;132(4):1183-90. doi: 10.1378/chest.07-0808. Epub 2007 Jul 23. PMID 17646221